CLINICAL TRIAL: NCT05072041
Title: Safety and Efficacy of Degradable Microsphere in Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma: a Prospective Comparative Study
Brief Title: Safety and Efficacy of Degradable Microsphere in Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEXTBIO-UIGB-HCC01
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group (Experimental): Degradable embolic microsphere (Nexsphere™)
  Interventions: Device: Nexsphere™

INTERVENTIONS:
Device: Nexsphere™ — Nexsphere™ is a yellow powder, made of 100% hydrophilic gelatin. It is used to make a suspension by mixing a contrast agent and physiological saline. The indications are hepatic artery chemoembolization, uterine artery embolization, prostate artery embolization, and treatment of various hemorrhagic diseases. It physically embolizes blood vessels and is decomposed within 4-8 weeks after intravascular injection.

SUMMARY:
The purpose of this study was to prospectively collect clinical data from patients who underwent hepatic artery chemoembolization using microspheres with different degradation times (2 hours, 1 day, 2 weeks) based on standard treatment.

DETAILED DESCRIPTION:
This study is a prospective study, and the purpose of this study is to investigate and collect clinical information on the safety and efficacy of degradable microsphere for hepatic artery chemoembolization in hepatocellular carcinoma patients. The primary purpose of this study was to evaluate the incidence of postembolism syndrome and liver function impairment after hepatic artery chemoembolization, and the secondary purpose was to evaluate tumor treatment response and hepatic artery damage after 1 month of hepatic artery chemoembolization.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 19 to 79 years
2. Patient who signed Informed Consent Form
3. Patients diagnosed with hepatocellular carcinoma by American Association for the Study of Liver Diseases (AASLD) and at least one of the following methods i. Magnetic resonance imaging (MRI) with early augmentation and delayed excretion of at least one solid liver lesion greater than 1 ㎝.

   ii. Contrast-enhanced computed tomography (CT) with early augmentation and delayed build-up of at least one solid liver lesion >1 ㎝.

   iii. Lesions with inconclusive features require histological confirmation.
4. Patients should not be eligible for treatment by amputation or percutaneous resection or liver transplantation at the time of study enrollment.

   i. Patients who are not suitable for ablation due to lesion location may be enrolled.

   ii. Patients with recurrent hepatocellular carcinoma who are not suitable for amputation or resection may be enrolled.
5. Must be Child-Pugh A or B hepatocellular carcinoma, and must satisfy the following criteria.

   i. Tumor lesion size from 1 ㎝ to 10 ㎝ ii. Number of tumors 1-7 iii. Physical activity European Cooperative Oncology Group (ECOG) ≤ 1 without vascular involvement
6. Patients who can be followed up until the end of the study and whose life expectancy is 6 months or longer

Exclusion Criteria:

1. Patients under the age of 19
2. Chronic kidney disease (CDK) grade 4 or 5 patients
3. Current or previous treatment with chemotherapy or radiation therapy or sorafenib or drug release chemoembolization (deTACE) after diagnosis of hepatocellular carcinoma

5. Pregnant, lactating, pre-menopausal and women not using effective contraceptive methods 6. Performance state European Cooperative Oncology Group (ECOG) > 1 7. Child-Poo Class C 8. Advanced hepatocellular carcinoma with vascular invasion or extrahepatic metastasis 9. Active Gastrointestinal Bleeding 10. Evidence of irreversible bleeding constitution 11. Encephalopathy that is not medically adequately controlled 12. Presence of ascites that is not medically controlled 13. Contraindications to Magnetic Resonance Imaging or Computed Tomography scan (e.g. metal implants) 14. Allergy to contrast media that cannot be managed by prevention 15. Contraindications to angiography 16. Contraindications to the administration of cisplatin anticancer drugs 17. Contraindications to hepatic artery embolization

* Extensive context-to-systemic shunts
* hepatofugal portal blood flow
* Serum bilirubin > 3.0 ㎎/dL
* Serum creatinine > 2.0 ㎎/dL
* Other symptoms that your doctor has determined to be exclusive.
* Irreversible blood clotting disorders 18. Others who are judged to be difficult for the principal investigator or principal investigator to conduct this clinical trial for other reasons

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postembolism syndrome | 8 weeks
  Nausea, vomiting, persistent pain, fever, and other
Incidence of liver function impairment | 8 weeks
  AFP, AST, ALT, BILI, GGT, BUN, and CREAT level

SECONDARY OUTCOMES:
Tumor treatment response | 8 weeks
  Evaluation of tumor size by Magnetic Resonance Imaging or Computed Tomography scan at 4 and 8 weeks after embolization
Hepatic artery damage | 8 weeks
  Vessel dissection, vessel stenosis, vessel occlusion, vessel wall irregularity, and other

CONTACTS AND LOCATIONS:
Overall Officials: Dong Il Gwon, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No